CLINICAL TRIAL: NCT00809770
Title: Contingency Management of Psychostimulant Abuse in the Severely Mentally Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard Ries, Director Division of Addiction, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDA022476A; R01DA022476 (NIH); R01DA022476-01 (NIH)
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Drug Abuse; Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: stimulant abuse; drug abuse; schizophrenia; bipolar disorder; major depressive disorder; contingency management; psychosocial treatment
MeSH Terms: conditions — Substance-Related Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Contingency management
  Interventions: Behavioral: Contingency Management
- 2 (Other): Non Contingent Control Condition
  Interventions: Behavioral: Non Contingent Control Condition

INTERVENTIONS:
Behavioral: Contingency Management — Opportunities to earn rewards are given three times a week for 12 weeks contingent on negative urine analyses indicating drug abstinence
  Arms: 1
Behavioral: Non Contingent Control Condition — Opportunities to draw for rewards are provided three times a week for 12 weeks for providing urine analysis. Opportunities to earn rewards are not based on urine analysis results.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness of a behavioral treatment, contingency management, in reducing stimulant use in persons with serious mental illness.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of a twelve week contingency management (CM) intervention for treating psycho-stimulant substance abuse when delivered in the context of a community mental health center (CMHC) setting for adults suffering from serious mental illness (SMI). The CM paradigm to be used is one which has been shown effective in several recent large clinical trials, using the variable magnitude of reinforcement procedure. The reinforcers will be vouchers or actual items useful for day to day living in this population. Two hundred SMI participants with co-occurring stimulant disorders will be recruited from a large urban CMHC and randomized to receive either the active CM paradigm plus treatment as usual (TAU), or TAU which will include the delivery of reinforcement for study involvement (reinforcement that is not contingent on drug abstinence). The primary outcome is change in psycho-stimulant use (methamphetamine, amphetamine and/or cocaine). Secondary outcomes include: changes in use of other illegal drugs or alcohol; changes in CMHC treatment adherence and follow-through; changes in psychiatric symptoms, quality of life, and community outcomes (homelessness, incarcerations, etc.). Additional outcomes to be measured include changes in drug craving, stage of change, nicotine use, and HIV risk status. The study involves two phases, the 12 week treatment phase, where CM and control treatments are delivered, as well as a 3 month follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patient at Community Psychiatric Clinic (CPC), a large mental health center in urban Seattle, Washington;
* Between 18 and 65 years of age;
* Diagnosis of of methamphetamine, amphetamine(illegal), or cocaine dependence or abuse;
* CPC medical record diagnosis of schizophrenia, schizoaffective disorder, bipolar I or II, or recurrent major depressive disorder
* Stimulant drug use one month before enrollment;
* Ability to understand written and spoken English;
* CPC clinical case manager must affirm the potential participant's ability to provide informed consent and clinical appropriateness (i.e., safety/severity of mental/substance/ physical health) to participate in the study.

Exclusion Criteria:

* Any medical/psychiatric condition, or severity of that condition, that, in the opinion of Dr. Ries, the PI, would compromise safe study participation
* Chart defined organic brain disorder or dementia;
* Current participation in a methadone maintenance program;
* Any other circumstances that in the PI's opinion precludes safe study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Stimulant drug use as measured by urine analysis | Treatment phase: 12 weeks (3 measurements a week), Follow Up Phase: 3 months (1 measuresment a month)

SECONDARY OUTCOMES:
Self report drug use | Measured monthly througout the study
Other drug use as measured by urine analysis | Treatment phase: 12 weeks (3 measurements a week), Follow Up Phase: 3 months (1 measuresment a month)
Symptoms of mental illness | Monthly throughout the study
Community outcomes (jail bookings, ER visits, mental health outcomes) | The entire study period and three months prior and after study involvement

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Ries, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Srebnik DS, McDonell MG, Ries RK, Andrus G. Conflicts among CMHC clinicians over the role of urine drug testing. Psychiatr Serv. 2014 May 1;65(5):700-1. doi: 10.1176/appi.ps.201300489. No abstract available. PMID 24788740
- [Derived] McDonell MG, Srebnik D, Angelo F, McPherson S, Lowe JM, Sugar A, Short RA, Roll JM, Ries RK. Randomized controlled trial of contingency management for stimulant use in community mental health patients with serious mental illness. Am J Psychiatry. 2013 Jan;170(1):94-101. doi: 10.1176/appi.ajp.2012.11121831. PMID 23138961